CLINICAL TRIAL: NCT04419493
Title: Bioequivalence of Alteplase Derived From Two Different Manufacturing Processes Following Intravenous Administration in Healthy Male Volunteers
Brief Title: A Study in Healthy Men to Compare 2 Different Formulations of Alteplase
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0135-0340; 2019-004932-40 (EudraCT Number)
Record Dates: First submitted 2020-06-04; First posted 2020-06-05 (Actual); Results first posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Healthy
MeSH Terms: interventions — Tissue Plasminogen Activator; Heparin

STUDY DESIGN:
Intervention Model Description: Part A: Open label Part B: Adaptive two-stage group-sequential design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part B: Alteplase, TPA-02 then Alteplase, TPA-05 (Experimental)
  Interventions: Drug: Alteplase (from modified manufacturing process); Drug: Heparin-Natrium-5000-ratiopharm (unfractionated heparin)
- Part B: Alteplase, TPA-05 then Alteplase, TPA-02 (Active Comparator)
  Interventions: Drug: Alteplase (from current manufacturing process); Drug: Heparin-Natrium-5000-ratiopharm (unfractionated heparin)
- Part A: Alteplase, TPA-05 then Alteplase, TPA-02 (Experimental): Open-label
  Interventions: Drug: Alteplase (from modified manufacturing process); Drug: Heparin-Natrium-5000-ratiopharm (unfractionated heparin)
- Part A: Alteplase, TPA-02 then Alteplase, TPA-05 (Active Comparator)
  Interventions: Drug: Alteplase (from current manufacturing process); Drug: Heparin-Natrium-5000-ratiopharm (unfractionated heparin)

INTERVENTIONS:
Drug: Alteplase (from modified manufacturing process) — Alteplase, TPA-05
  Arms: Part A: Alteplase, TPA-05 then Alteplase, TPA-02; Part B: Alteplase, TPA-02 then Alteplase, TPA-05
Drug: Alteplase (from current manufacturing process) — Alteplase, TPA-02
  Arms: Part A: Alteplase, TPA-02 then Alteplase, TPA-05; Part B: Alteplase, TPA-05 then Alteplase, TPA-02
Drug: Heparin-Natrium-5000-ratiopharm (unfractionated heparin) — Heparin-Natrium-5000-ratiopharm (unfractionated heparin)

SUMMARY:
To establish the bioequivalence of alteplase derived from two different manufacturing processes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 45 years (inclusive)
* Body mass index (weight divided by height squared) (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Body weight of 65 - 100 kg (inclusive) at screening
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance, e.g. thrombotic predisposition according to thrombophilic testing
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity
* During COVID-19 pandemic: laboratory test indicative of an ongoing SARS-CoV-2 infection Further exclusion criteria apply.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Glund S, Hoefler J, Lang B, Cafiero S, Panova-Noeva M, Place C, Wolff M. Bioequivalence of Intravenous Alteplase from Two Different Manufacturing Processes in Healthy Male Volunteers: Results from a Two-Stage, Adaptive-Design Study. Clin Pharmacokinet. 2023 Jul;62(7):1023-1030. doi: 10.1007/s40262-023-01253-3. Epub 2023 May 30. PMID 37248330
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomised, open-label, 2 -way cross-over design with at least 24 h wash-out, to establish the bioequivalence of alteplase derived from two different manufacturing processes (new process, tissue plasminogen activator (TPA)-05, vs. current process, TPA-02) in healthy male volunteers.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated. In this cross-over trial 2 single doses of alteplase were infused on 2 consecutive days keeping a wash-out period of at least 24 h.
Groups:
- Part A: Alteplase, TPA-02 Then Alteplase, TPA-05: Participants were administered on Day 1 of Period 1 a single dose of 0.2 milligram (mg)/kilogram (kg) body weight of alteplase from current manufacturing process (alteplase, TPA-02) intravenously (i.v.) over a 30 minutes (min) infusion.
  On Day 1 of Period 2 participants were administered a single dose of 0.2 mg/kg body weight of alteplase from modified manufacturing process (alteplase, TPA-05) intravenously (i.v.) over a 30 min infusion.
  The 2 treatment periods were separated by a washout period of at least 24 hours (h).
- Part A: Alteplase, TPA-05 Then Alteplase, TPA-02: Participants were administered on Day 1 of Period 1 a single dose of 0.2 milligram (mg)/kilogram (kg) body weight of alteplase from modified manufacturing process (alteplase, TPA-05) intravenously (i.v.) over a 30 minutes (min) infusion.
  On Day 1 of Period 2 participants were administered a single dose of 0.2 mg/kg body weight of alteplase from current manufacturing process (alteplase, TPA-02) intravenously (i.v.) over a 30 min infusion.
  The 2 treatment periods were separated by a washout period of at least 24 hours (h).
- Part B: Alteplase, TPA-02 Then Alteplase, TPA-05: Participants were administered on Day 1 of Period 1 a single dose of 0.2 milligram (mg)/kilogram (kg) body weight of alteplase from current manufacturing process (alteplase, TPA-02) intravenously (i.v.) over a 30 minutes (min) infusion. 5 min prior to the infusion of alteplase, TPA-02, participants were administered 5000 international units (IU) of the auxiliary medicinal product (AMP) unfractionated heparin (Heparin-Natrium-ratiopharm®) as an intravenous bolus.
  On Day 1 of Period 2 participants were administered a single dose of 0.2 mg/kg body weight of alteplase from modified manufacturing process (alteplase, TPA-05) intravenously (i.v.) over a 30 min infusion. 5 min prior to the infusion of alteplase, TPA-05, participants were administered 5000 international units (IU) of the auxiliary medicinal product (AMP) unfractionated heparin (Heparin-Natrium-ratiopharm®) as an intravenous bolus.
  The 2 treatment periods were separated by a washout period of at least 24 hours (h).
- Part B: Alteplase, TPA-05 Then Alteplase, TPA-02: Participants were administered on Day 1 of Period 1 a single dose of 0.2 milligram (mg)/kilogram (kg) body weight of alteplase from modified manufacturing process (alteplase, TPA-05) intravenously (i.v.) over a 30 minutes (min) infusion. 5 min prior to the infusion of alteplase, TPA-05, participants were administered 5000 international units (IU) of the auxiliary medicinal product (AMP) unfractionated heparin (Heparin-Natrium-ratiopharm®) as an intravenous bolus.
  On Day 1 of Period 2 participants were administered a single dose of 0.2 mg/kg body weight of alteplase from current manufacturing process (alteplase, TPA-02) intravenously (i.v.) over a 30 min infusion. 5 min prior to the infusion of alteplase, TPA-02, participants were administered 5000 international units (IU) of the auxiliary medicinal product (AMP) unfractionated heparin (Heparin-Natrium-ratiopharm®) as an intravenous bolus.
  The 2 treatment periods were separated by a washout period of at least 24 hours (h).
Period: Period 1
Arm/Group | Part A: Alteplase, TPA-02 Then Alteplase, TPA-05 | Part A: Alteplase, TPA-05 Then Alteplase, TPA-02 | Part B: Alteplase, TPA-02 Then Alteplase, TPA-05 | Part B: Alteplase, TPA-05 Then Alteplase, TPA-02
Started | 6 | 6 | 9 | 9
Completed | 6 | 6 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Wash-out After Period 1
Arm/Group | Part A: Alteplase, TPA-02 Then Alteplase, TPA-05 | Part A: Alteplase, TPA-05 Then Alteplase, TPA-02 | Part B: Alteplase, TPA-02 Then Alteplase, TPA-05 | Part B: Alteplase, TPA-05 Then Alteplase, TPA-02
Started | 6 | 6 | 9 | 9
Completed | 5 | 4 | 8 | 9
Not Completed | 1 | 2 | 1 | 0
Not completed — Adverse Event | 1 | 2 | 1 | 0
Period: Period 2
Arm/Group | Part A: Alteplase, TPA-02 Then Alteplase, TPA-05 | Part A: Alteplase, TPA-05 Then Alteplase, TPA-02 | Part B: Alteplase, TPA-02 Then Alteplase, TPA-05 | Part B: Alteplase, TPA-05 Then Alteplase, TPA-02
Started | 5 | 4 | 8 | 9
Completed | 5 | 4 | 8 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set - part A (TS-A) included all subjects who were randomised and treated with at least 1 dose of the investigational medicinal product.
  Treated set - part B (TS-B) included all subjects who had been randomised and treated with at least 1 dose of the investigational medicinal product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Alteplase, TPA-02 Then Alteplase, TPA-05 | Part A: Alteplase, TPA-05 Then Alteplase, TPA-02 | Part B: Alteplase, TPA-02 Then Alteplase, TPA-05 | Part B: Alteplase, TPA-05 Then Alteplase, TPA-02 | Total
Number analyzed (Participants) | 6 | 6 | 9 | 9 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.3 (5.8) | 32.2 (6.2) | 31.7 (5.8) | 35.8 (5.8) | 33.5 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 9 | 9 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 6 | 9 | 8 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 6 | 6 | 9 | 8 | 29
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Area Under the Concentration-time Curve of Alteplase in Plasma Over the Time Interval From 0 up to the Last Quantifiable Data Point (AUC0-tz)
Description: The area under the concentration-time curve of alteplase in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) is reported.
Time Frame: Within 3 hours (h) before and 5 minutes (min), 10min, 15min, 20min, 25min, 30min, 32min, 34min, 36min, 40min, 45min, 50min, 1h, 1.33h, 1.67h, 2h, 3h, 4h and 6h after start of alteplase infusion.
Population: Pharmacokinetic parameter analysis set - part A (PKS-A): Includes all subjects in the treated set - part A (TS-A) who provide at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol violation to the evaluation of PK or due to PK non-evaluability. PK data for Part A were not used for the final assessment of bioequivalence according to protocol amendment after obtaining unreliable PK results.
Groups:
- Part A: Alteplase, TPA -02: Participants were administered during trial Part A a single dose of 0.2 milligram (mg)/kilogram (kg) body weight of alteplase from current manufacturing process (alteplase, TPA-02) intravenously (i.v.) over a 30 minutes (min) infusion.
- Part A: Alteplase, TPA-05: Participants were administered during trial Part B a single dose of 0.2 milligram (mg)/kilogram (kg) body weight of alteplase from modified manufacturing process (alteplase, TPA-05) intravenously (i.v.) over a 30 minutes (min) infusion.
Arm/Group | Part A: Alteplase, TPA -02 | Part A: Alteplase, TPA-05
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Part B: Area Under the Concentration-time Curve of Alteplase in Plasma Over the Time Interval From 0 up to the Last Quantifiable Data Point (AUC0-tz)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter analysis set - part B(PKS-B): This set includes all subjects in the treated set - part B (TS-B) who provide at least one Pharmacokinetic (PK) endpoint that was defined as primary or secondary and was not excluded due to a protocol violation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Least Squares Mean (Standard Error); unit: hour * nanogram / milliliter (h*ng/mL)
Groups:
- Part B: Alteplase, TPA -02: Participants were administered during trial Part B a single dose of 0.2 milligram (mg)/kilogram (kg) body weight of alteplase from current manufacturing process (alteplase, TPA-02) intravenously (i.v.) over a 30 minutes (min) infusion. 5 min prior to the infusion of alteplase, TPA-02, participants were administered 5000 international units (IU) of the auxiliary medicinal product (AMP) unfractionated heparin (Heparin-Natrium-ratiopharm®) as an intravenous bolus.
- Part B: Alteplase, TPA-05: Participants were administered during trial Part B a single dose of 0.2 milligram (mg)/kilogram (kg) body weight of alteplase from modified manufacturing process (alteplase, TPA-05) intravenously (i.v.) over a 30 minutes (min) infusion. 5 min prior to the infusion of alteplase, TPA-05, participants were administered 5000 international units (IU) of the auxiliary medicinal product (AMP) unfractionated heparin (Heparin-Natrium-ratiopharm®) as an intravenous bolus.
Arm/Group | Part B: Alteplase, TPA -02 | Part B: Alteplase, TPA-05
Number analyzed (Participants) | 16 | 16
hour * nanogram / milliliter (h*ng/mL) | 369.21 (NA) — The standard error is actually adjusted standard error and is equal to 1.03. | 377.35 (NA) — The standard error is actually adjusted standard error and is equal to 1.03.
Statistical Analysis 1: Comparison: Part B: Alteplase, TPA -02 vs Part B: Alteplase, TPA-05; The null hypothesis was that the ratio of expected geometric least squares means Alteplase, TPA-02 vs. Alteplase, TPA-05 is less than 80.00% or more than 125.00%. The statistical model used for the analysis of this endpoints was an analysis of variance (ANOVA) model on the logarithmic scale. This model included effects accounting for the following sources of variation: sequence, subjects within sequences, period and treatment. All effects were considered as fixed; Test type: Equivalence — Bioequivalence was concluded, if the confidence interval (CI) for the comparison of geometric least squares means ratio was included in the pre-defined equivalence range of 80.00% to 125.00%; Geometric Least Squares Mean ratio (%) = 102.20, 92.83% CI 2-sided [94.87 to 110.10], Standard Error of Mean 10.8 — Geometric Least Squares Mean ratio is: Alteplase, TPA-02/Alteplase, TPA-05. Standard Error of the mean is actually the intra-individual geometric coefficient variation

3. Primary Outcome: Part A: Maximum Measured Concentration of Alteplase in Plasma (Cmax)
Description: Maximum measured concentration of alteplase in plasma is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Groups:
- Part A: Alteplase, TPA-05: Participants were administered during trial Part A a single dose of 0.2 milligram (mg)/kilogram (kg) body weight of alteplase from modified manufacturing process (alteplase, TPA-05) intravenously (i.v.) over a 30 minutes (min) infusion.
Arm/Group | Part A: Alteplase, TPA -02 | Part A: Alteplase, TPA-05
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Part B: Maximum Measured Concentration of Alteplase in Plasma (Cmax)
Description: Maximum measured concentration of Alteplase in plasma (Cmax) is reported.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Least Squares Mean (Standard Error); unit: nanogram / milliliter (ng/mL)
Arm/Group | Part B: Alteplase, TPA -02 | Part B: Alteplase, TPA-05
Number analyzed (Participants) | 16 | 16
nanogram / milliliter (ng/mL) | 738.35 (NA) — The standard error is actually adjusted standard error and is equal to 1.02. | 781.24 (NA) — The standard error is actually adjusted standard error and is equal to 1.02.
Statistical Analysis 1: Comparison: Part B: Alteplase, TPA -02 vs Part B: Alteplase, TPA-05; [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Least Squares Mean ratio (%) = 105.81, 92.83% CI 2-sided [99.18 to 112.88], Standard Error of Mean 9.3 — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Part A: Area Under the Concentration-time Curve of Alteplase in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of alteplase in plasma over interval from 0 extrapolated to infinity is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Part A: Alteplase, TPA -02 | Part A: Alteplase, TPA-05
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Part B: Area Under the Concentration-time Curve of Alteplase in Plasma Over the Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of alteplase in plasma over the interval from 0 extrapolated to infinity is reported.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*nanogram/milliliter (h*ng/mL)
Arm/Group | Part B: Alteplase, TPA -02 | Part B: Alteplase, TPA-05
Number analyzed (Participants) | 16 | 16
hour*nanogram/milliliter (h*ng/mL) | 371.85 (NA) — The standard error is actually adjusted standard error and is equal to 1.03. | 379.90 (NA) — The standard error is actually adjusted standard error and is equal to 1.03.
Statistical Analysis 1: Comparison: Part B: Alteplase, TPA -02 vs Part B: Alteplase, TPA-05; [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — Bioequivalence was concluded, if the confidence interval (CI) for the comparison of geometric least squares means ratio was included in the pre-defined equivalence range of 80.00% to 125.00%; Geometric Least Squares Mean ratio (%) = 102.17, 92.83% CI 2-sided [94.79 to 110.12], Standard Error of Mean 10.8 — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to 22 days after the last administration of alteplase.
Description: Treated set - part A (TS-A) and Treated set - part B (TS-B): The treated sets includes all subjects who were randomized and treated with at least one dose of study drug.
Groups:
- Part A: Alteplase, TPA-02: Participants were administered during trial Part A a single dose of 0.2 milligram (mg)/kilogram (kg) body weight of alteplase from current manufacturing process (alteplase, TPA-02) intravenously (i.v.) over a 30 minutes (min) infusion.
- Part B: Alteplase, TPA-02: Participants were administered during trial Part B a single dose of 0.2 milligram (mg)/kilogram (kg) body weight of alteplase from current manufacturing process (alteplase, TPA-02) intravenously (i.v.) over a 30 minutes (min) infusion. 5 min prior to the infusion of alteplase, TPA-02, participants were administered 5000 international units (IU) of the auxiliary medicinal product (AMP) unfractionated heparin (Heparin-Natrium-ratiopharm®) as an intravenous bolus.
Arm/Group | Part A: Alteplase, TPA-02 | Part B: Alteplase, TPA-02 | Part A: Alteplase, TPA-05 | Part B: Alteplase, TPA-05
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/18 | 0/11 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/18 | 0/11 | 0/17
Other Adverse Events (participants affected / at risk) | 1/10 | 7/18 | 4/11 | 6/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Alteplase, TPA-02 (N=10) | Part B: Alteplase, TPA-02 (N=18) | Part A: Alteplase, TPA-05 (N=11) | Part B: Alteplase, TPA-05 (N=17)
Catheter site paraesthesia (General disorders) | 0 | 0 | 1 | 0
Catheter site swelling (General disorders) | 0 | 1 | 1 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1 | 1
Catheter site haematoma (General disorders) | 0 | 0 | 0 | 2
Catheter site pain (General disorders) | 0 | 2 | 0 | 0
Infusion site pain (General disorders) | 0 | 1 | 0 | 1
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Device occlusion (Product Issues) | 1 | 0 | 2 | 1

LIMITATIONS AND CAVEATS:
For study Part A three subjects underwent only one treatment period, thereafter the trial was put on-hold. Trial Part B was performed as planned. There were no important protocol deviations (IPDs). Each entered subject met all of the inclusion criteria and none of the exclusion criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT04419493/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT04419493/SAP_001.pdf